CLINICAL TRIAL: NCT01064128
Title: Randomized Controlled Study of Different Pain Scores in Single-Port Access (SPA) Laparoscopic Hysterectomy Versus Conventional Laparoscopic Hysterectomy
Brief Title: Study of Different Pain Scores in Single-Port Access (SPA) Laparoscopic Hysterectomy Versus Conventional Laparoscopic Hysterectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Tae Joong, Kim/Clinical Assistant Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-09-093
Record Dates: First submitted 2010-02-05; First posted 2010-02-08 (Estimated); Last update posted 2011-07-20 (Estimated); Status verified 2011-07

CONDITIONS: Uterine Myoma; Uterine Adenomyosis
Keywords: Single-port; Laparoscopy; Hysterectomy; Pain; Cosmesis; Analgesics
MeSH Terms: conditions — Myofibroma; Adenomyosis; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- conventional laparoscopic hysterectomy (Active Comparator): Three or four ports conventional laparoscopic hysterectomy
  Interventions: Procedure: conventional laparoscopic hysterectomy
- SPA laparoscopic hysterectomy (Active Comparator): Single umbilical incision laparoscopic hysterectomy
  Interventions: Procedure: SPA laparoscopic hysterectomy

INTERVENTIONS:
Procedure: conventional laparoscopic hysterectomy — conventional 3 or 4 ports laparoscopic hysterectomy
  Arms: conventional laparoscopic hysterectomy
Procedure: SPA laparoscopic hysterectomy — single-port access laparoscopic hysterectomy
  Arms: SPA laparoscopic hysterectomy

SUMMARY:
Purpose:

The attempt to further reduce the operative trauma in laparoscopic hysterectomy led in new technique such as Single-Port Access (SPA) laparoscopic surgery. This new technique is considered as painless procedure and better cosmetic effect but there are not any publications to study a possible different pain score and cosmetic effect in new techniques versus conventional laparoscopic hysterectomy. In this randomized controlled study the researchers have investigated the pain scores and cosmetic satisfaction by modified body image scale and cosmetic scar scale.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-60, female
* Symptomatic (Dysmenorrhea, Palpable mass, Pelvic pain or discomfort, Urinary symptom, Increasing size, Menorrhagia) myomas or adenomyosis
* Suspected uterine myoma and/or adenomyosis on transvaginal ultrasonography (USG)
* At least a 6-month thorough follow-up record available
* Informed consent

Exclusion Criteria:

* Endometrial hyperplasia without myoma or adenomyosis
* Body Mass Index more than 30
* Huge uterus defined by longitudinal uterine diameter larger than 10cm and anteroposterior diameter larger than 8cm in USG

Ages: 30 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Pain score measured by visual analog scale | postoperative 24 hours

SECONDARY OUTCOMES:
Modified body image scale and cosmetic scar scale | postoperative 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea